CLINICAL TRIAL: NCT04995068
Title: Stockholm Score of Lesion Development on Computerized Tomography Following Mild Traumatic Brain Injury
Brief Title: Score Predicting Lesion Development on CT Following Mild TBI
Acronym: SELECT-TBI
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); St Goran's Hospital (Other); Norrtalje Hospital (Unknown); Danderyd Hospital (Other); Sodertalje Hospital (Other)
Responsible Party: Principal Investigator, Eric Thelin, Principle Investigator, Karolinska Institutet
Other Study IDs: 2020-05728
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury
Keywords: neurosurgery
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Included patients: See inclusion and exclusion criteria
  Interventions: Radiation: Head CT to determine presence of traumatic intracranial lesion

INTERVENTIONS:
Radiation: Head CT to determine presence of traumatic intracranial lesion — Head CT to determine presence of traumatic intracranial lesion

SUMMARY:
Mild traumatic brain injury (mTBI) is one of the most common reasons behind emergency department (ED) visits. A small portion of mTBI patients will develop an intracranial lesion that might require neurosurgical intervention. Several guidelines have been developed to help direct these patients for head Computerized Tomography (CT) scanning, but they lack specificity, mainly focus on ruling out lesions, and do not estimate the risk of lesion development. The aim of this retrospective observational study is to create a risk stratification score that predicts the likelihood of intracranial lesion development, lesion progression, and need for neurosurgical management in patients with mTBI presenting to the ED. Eligible patients are adults (≥ 15 years) with mTBI (defined as admission Glasgow Coma Scale (GCS) 13-15) who presented to the ED within 24 hours of injury to any ED in Stockholm, Sweden between 2010-2020. Reasons for ED visit and Internal Classification of Disease (ICD) codes will be used to screen for patients. Machine-learning models will be applied. The primary outcome will be a traumatic lesion on head CT, defined as a cerebral contusion, subdural haematoma, epidural haematoma, subarachnoid haemorrhage, intraventricular haemorrhage, diffuse axonal injury, skull fracture, traumatic infarction or sinus thrombosis. The secondary outcomes will be any clinically significant lesion, defined as an intracranial finding that led to neurosurgical intervention, discontinuation or reversal of anticoagulant or antiplatelet medication, hospital admission > 48 hours due to the TBI, or death.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 15 years)
* Presented to emergency department within 24 hours of TBI
* GCS 13-15 at presentation to the emergency department

Exclusion Criteria:

* No CT scan performed
* Patient from another Region in Sweden/another country
* Penetrating TBI
* Secondary transfer from other emergency department
* Medical record missing

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (≥ 15 years) with mild traumatic brain injury (GCS 13-15) who presented to the emergency department within 24 hours of injury.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Traumatic intracranial lesion | Immediately after the procedure (CT-scan)
  Any traumatic lesion on head CT, defined as a cerebral contusion, subdural haematoma, epidural haematoma, subarachnoid haemorrhage, intraventricular haemorrhage, diffuse axonal injury, skull fracture, traumatic infarction or sinus thrombosis.

SECONDARY OUTCOMES:
Clinically significant traumatic intracranial lesion | Immediately after the procedure (CT-scan)
  Primary outcome measure that led to neurosurgical intervention, discontinuation or reversal of anticoagulant or antiplatelet medication, hospital admission > 48 hours due to the TBI, or death due to TBI
Lesion progression | Within 48 hours of the first CT-scan
  Hemorrhagic primary outcome measure (cerebral contusion, subdural haematoma, epidural haematoma, subarachnoid haemorrhage or intraventricular haemorrhage) that progressed on a follow-up CT

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Thelin, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the planned study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Following publication of the study, the above will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Yang LJ, Tatter C, Fletcher-Sandersjoo A, Froese L, Lassaren P, Tjerkaski J, Bergman EE, Bjorkman FE, Bronge J, Antonsson J, Teromaa K, Nylander M, Ortqvist S, Kylander W, Lindqvist W, Angeby K, Rubenson Wahlin R, Thelin EP. Stockholm Score of Lesion Detection on Computed Tomography following Mild Traumatic Brain Injury (SELECT-TBI) Study: Pilot Analysis and Statistical Analysis Plan. Acta Neurochir (Wien). 2025 Jul 1;167(1):181. doi: 10.1007/s00701-025-06598-1. PMID 40591064
- [Derived] Fletcher-Sandersjoo A, Tatter C, Yang L, Ponten E, Boman M, Lassaren P, Forsberg S, Gronlund I, Tidehag V, Rubenson-Wahlin R, Strommer L, Westberg K, Angeby K, Djarv T, Lundblad O, Bartek J Jr, Thelin EP. Stockholm score of lesion detection on computed tomography following mild traumatic brain injury (SELECT-TBI): study protocol for a multicentre, retrospective, observational cohort study. BMJ Open. 2022 Sep 1;12(9):e060679. doi: 10.1136/bmjopen-2021-060679. PMID 36581962